CLINICAL TRIAL: NCT03619694
Title: Role of Magnetic Resonance Spectroscopy in Differentiating Brain Tumors
Brief Title: Role of MR Spectroscopy in Brain Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelwahab, Principal investigator, Assiut University
Other Study IDs: MRS in brain tumors
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Brain Neoplasms
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI Spectroscopy — Patient with brain SOL underwent MRI Spectroscopy to be compared with later pathology

SUMMARY:
In order to come as close as possible to the correct diagnosis of CNS tumors, MRI is the long-standing accepted method of choice that can in some cases be supported by the use of CT to demonstrate calcification or bone destruction. In individual cases MRI spectroscopy can be helpful for the differentiation between neoplasms and inflammatory lesions or surveillance of tumor therapy, just as perfusion

DETAILED DESCRIPTION:
Proton magnetic resonance spectroscopy (H-MRS) may be helpful in suggesting tumor histology and tumor grade and may better define tumor extension and the ideal site for biopsy compared with conventional magnetic resonance (MR) imaging. A multifunctional approach with diffusion-weighted imaging, perfusion-weighted imaging, and permeability maps, along with H-MRS, may enhance the accuracy of the diagnosis and characterization of brain tumors and estimation of therapeutic response. Integration of advanced imaging techniques with conventional MR imaging and the clinical history help to improve the accuracy, sensitivity, and specificity in differentiating tumors and nonneoplastic lesions.

ELIGIBILITY:
Inclusion Criteria:

* All patients with space-occupying lesions

Exclusion Criteria:

* Post operative cases
* Non-neoplastic nature

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with brain tumors diagnosed by conventional imaging
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of MRS findings with the pathology of the specimens | Baseline
  Analysis of the MRS metabolites peaks and integral and test if they can differentiate the grades of brain tumors

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Peitgen N, Papanagiotou P. [Intra-axial brain tumors in adults : On the basis of the 2016 WHO classification]. Radiologe. 2017 Sep;57(9):707-714. doi: 10.1007/s00117-017-0271-6. German. PMID 28667395
- [Background] Brindle KM, Izquierdo-Garcia JL, Lewis DY, Mair RJ, Wright AJ. Brain Tumor Imaging. J Clin Oncol. 2017 Jul 20;35(21):2432-2438. doi: 10.1200/JCO.2017.72.7636. Epub 2017 Jun 22. PMID 28640699